CLINICAL TRIAL: NCT07256002
Title: Survival Analysis and Prognostic Biomarker Exploration of Postoperative Adjuvant Therapy Patterns in Patients With Non-small Cell Lung Cancer After Neoadjuvant Immunotherapy:A Real World Multicenter Retrospective Study
Brief Title: Survival Analysis and Prognostic Biomarker Exploration of Postoperative Adjuvant Therapy Patterns in Patients With Non-small Cell Lung Cancer After Neoadjuvant Immunotherapy
Status: Active, not recruiting | Type: Observational
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: NCC5704
Record Dates: First submitted 2025-09-28; First posted 2025-12-01 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-09

CONDITIONS: Lung Cancer (NSCLC)
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Immune Checkpoint Inhibitors; Drug Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: PD-1 Inhibitors — Adjuvant PD-1 inhibitor maintenance therapy
Drug: Chemotherapy — Postoperative chemotherapy as an adjuvant treatment
Drug: PD-1 inhibitors combined with chemotherapy — Postoperative PD-1 inhibitor combined with chemotherapy as adjuvant therapy

SUMMARY:
The aim of this observational study is to investigate the survival differences among patients with non-small cell lung cancer who received different adjuvant treatments after neoadjuvant immunotherapy, and to identify the main clinical characteristics of these survival differences. The main question it aims to answer is:

1. Is there a difference in survival between patients who achieve pCR after neoadjuvant immunotherapy and those who do not receive adjuvant therapy?
2. What are the recurrence patterns and high-risk factors for recurrence in patients with pCR after neoadjuvant immunotherapy, and how can early intervention be carried out?
3. Is there a difference in survival among patients with non-MPR after neoadjuvant immunotherapy when they receive different adjuvant treatment modalities (single immunotherapy, chemio-immunotherapy, chemotherapy, etc.)?
4. Should patients with non-MPR after neoadjuvant immunotherapy continue immunotherapy, and what are the predictive markers for receiving adjuvant therapy?

DETAILED DESCRIPTION:
The aim of this observational study is to investigate the survival differences among patients with non-small cell lung cancer who received different adjuvant treatments after neoadjuvant immunotherapy, and to identify the main clinical characteristics of these survival differences. The main question it aims to answer is:

1. Is there a difference in survival between patients who achieve pCR after neoadjuvant immunotherapy and those who do not receive adjuvant therapy?
2. What are the recurrence patterns and high-risk factors for recurrence in patients with pCR after neoadjuvant immunotherapy, and how can early intervention be carried out?
3. Is there a difference in survival among patients with non-MPR after neoadjuvant immunotherapy when they receive different adjuvant treatment modalities (single immunotherapy, chemio-immunotherapy, chemotherapy, etc.)?
4. Should patients with non-MPR after neoadjuvant immunotherapy continue immunotherapy, and what are the predictive markers for receiving adjuvant therapy? Participants will undergo neoadjuvant immunotherapy and surgical procedures, and through rigorous analysis of real-world data, this study endeavors to provide nuanced insights into these fundamental queries, fostering advancements in clinical decision-making and patient management strategies.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who visited the hospital from January 2020 to December 2023;
2. Received neoadjuvant immunotherapy before surgery;
3. Histologically diagnosed with stage II-III NSCLC;
4. Had measurable lesions as assessed by the investigator using the RECIST 1.1 version;
5. Underwent radical surgical treatment;
6. ECOG score of 0 or 1;
7. Available tumor tissue samples;
8. Good blood and organ functions.

Exclusion Criteria:

1. Has received other anti-tumor treatments before, including radiotherapy, chemotherapy and traditional Chinese medicine-based cancer treatment (except for malignant tumor treatments that have been cured and have no recurrence or metastasis for more than 5 years);
2. Has a history of previous malignant tumors.

Ages: 18 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with lung cancer who have received neoadjuvant immunotherapy and surgery.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) | From date of diagnosis until the date of death from any cause, whichever came first, assessed up to 7 years and 11 months.
  OS is defined as the time from surgery time until death from any cause.

SECONDARY OUTCOMES:
Event-free survival(EFS) | up to 7 years and 11 months.
  Event-free survival was defined as the time from neoadjuvant treatment to metastasis or death by any cause in the absence of metastasis.
Pathological Complete Response(pCR) | up to 1 month after surgery
  After evaluating the removed tumor tissue and the regional lymph nodes, no residual tumor cells were found.

CONTACTS AND LOCATIONS:
Overall Officials: Shugeng Gao, MD, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (1):
- Cancer Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China